CLINICAL TRIAL: NCT05802641
Title: Clinical Study of Stereotactic Radiotherapy With Different Fractionation Modes for Early Lung Cancer
Brief Title: Stereotactic Radiotherapy With Different Fractionation Modes for the Early Lung Cancer
Acronym: DSBRT-1
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: DSBRT-1
Record Dates: First submitted 2023-03-26; First posted 2023-04-06 (Actual); Last update posted 2023-04-06 (Actual); Status verified 2023-03

CONDITIONS: Lung Cancer; Radiotherapy; Stereotactic Body Radiotherapy; Fractionation
Keywords: lung cancer; Stereotactic body radiotherapy; Fractionation
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- single fraction of SBRT（30Gy/1f）: Participants with early lung cancer receive single fraction of SBRT（30Gy/1f).
  Interventions: Radiation: SBRT
- Multiple fractions of SBRT（36Gy/3f）: Participants with early lung cancer receive multiple fractions of SBRT（36Gy/3f).
  Interventions: Radiation: SBRT

INTERVENTIONS:
Radiation: SBRT — Participants with early lung cancer receive single fraction (30Gy/1f) or multiple fractions of SBRT（36Gy/3f).

SUMMARY:
The goal of this observational study is to study the efficacy and safety of stereotactic body radiotherapy (SBRT) with different fractionation modes for early lung cancer. The main questions it aims to answer are:

How effective are different regimens of SBRT for early lung cancer? How safe are different regimens of SBRT of SBRT for early lung cancer?

DETAILED DESCRIPTION:
The goal of this observational study is to study the efficacy and safety of stereotactic body radiotherapy (SBRT) with different fractionation modes for early lung cancer.. This study intends to review the patients with early lung cancer receiving SBRT of 30Gy/1f or 36Gy/3f from 2018 to 2024 in our center.

ELIGIBILITY:
Inclusion Criteria:

1. Signed written informed consent;
2. Male or female aged ≥ 18 years and ≤ 75 years;
3. patients with early lung cancer confirmed by pathology or clinical multidisciplinary team (MDT);
4. The ECOG PS was 0 to 1;
5. Survival time ≥3 months;
6. Laboratory results during screening must meet the following requirements:

   1. Blood routine: neutrophil absolute count (ANC) ≥ 1.5 × 109/L, platelet count (PLT) ≥ 100 × 109/L, hemoglobin (HGB) ≥ 90 g/L (no blood transfusion or erythropoietin dependence within 7 days);
   2. Liver function: total bilirubin (TBIL) ≤ 1.5 times the upper limit of normal value (ULN); Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) were less than 2.5 times ULN in subjects without liver metastasis, and ALT and AST were less than 5 times ULN in subjects with liver metastasis.
   3. Renal function: serum creatinine (Cr) ≤1.5 times ULN or Cr clearance ≥60 mL/min (Cockcroft-Gault formula), and urine protein (UPRO) &lt on routine urine test; 2+ or 24 h urinary protein quantification < 1g;
   4. International standardized ratio (INR) ≤1.5 times ULN and partial prothrombin time (PTT) or activated partial thrombin time (APTT) ≤1.5 times ULN during the 7 days prior to treatment;

Exclusion Criteria:

1. any unstable systemic disease, including but not limited to active infection, congestive heart failure [New York Heart Association (NYHA) class ≥ II], severe arrhythmia requiring medical therapy, liver, kidney, or metabolic disease; Type I and type II respiratory failure;
2. other malignancies within 5 years before randomization, except adequately treated cervical carcinoma in situ, basal cell or squamous skin cancer, local prostate cancer after radical surgery, ductal carcinoma in situ after radical surgery, or papillary thyroid cancer;

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: This study intends to review the patients with early lung cancer receiving SBRT of 30Gy/1f or 36Gy/3f from 2018 to 2024 in our center.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2018-01-07 (Actual); Primary Completion 2024-01 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
PFS | 2025-01-01
  The time from the date of treatment to the date of disease progression or death or last follow-up.

SECONDARY OUTCOMES:
OS | 2025-01-01
  The time from the date of treatment to the date of death or last follow-up.
AE | 2025-03-21
  The incidence of All adverse event (AE), treatment emergent AE (TEAE), treatment-related AE (TRAE), serious AE (SAE) and radiation-related AE(rAE), the relevance and severity related with the study protocol.

CONTACTS AND LOCATIONS:
Overall Officials: Hongqing Zhuang, M.D., Principal Investigator — Department of Peking University Third Hospital
Locations (1):
- Department of radiation oncology, Peking University Third Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
Study Protocol, Statistical Analysis Plan, and Clinical Study Report will be shared with researchers for research use after permission was obtained from the study institution.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: starting 6 months after publication
Access Criteria: Only for researchers.